CLINICAL TRIAL: NCT06177353
Title: Etude du Profil Immunologique Sanguin et cutané Des Patients Atteints d'épidermolyse Bulleuse Dystrophique récessive : Analyses in Vivo et Impact Des Cellules Souches Placentaires in Vitro
Brief Title: Study of the Blood and Skin Immunological Profile of Patients With Recessive Dystrophic Epidermolysis Bullosa: in Vivo Analysis and the Impact of Placental Stem Cells in Vitro
Acronym: ISTRADEB
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230933
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Epidermolysis Bullosa Dystrophica
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EBDR patients
  Interventions: Other: Sampling
- Healthy control
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Blood sampling Skin biopsy Collection of soiled bandages

SUMMARY:
Patients with recessive dystrophic epidermolysis bullosa (RDEB) suffer from acute and chronic post-bullous wounds along with impaired skin healing. These issues are attributed not only to mucocutaneous fragility and abnormal healing directly related to quantitative and/or qualitative constitutional abnormalities of collagen VII but also to a contingent cutaneous and systemic inflammatory component. This inflammatory aspect contributes to the perpetuation of skin lesions and delayed healing. Our primary objective is to define the systemic immunological/inflammatory signature of patients with RDEB with an aim to develop a strategy that involves using stem cells with high immunomodulatory/anti-inflammatory capacity such as allogeneic placental stem cells (WJ-MSCs and trophoblasts).

ELIGIBILITY:
Inclusion Criteria:

EBDR patients :

* Patients aged 18 to 80 years old
* Clinically, histologically, and/or genetically confirmed intermediate, reversed or generalized, moderate to severe EBDR

Healthy controls :

* Adults aged 18 to 80 years old
* PBMC healthy donors: subjects who have donated blood to the EFS according to the indication criteria who have consented to the use of their samples for research purposes.
* Healthy skin biopsy donors: subjects undergoing abdominoplasty scheduled in plastic surgery and who have given their consent for the collection of a skin biopsy from post-operative abdominoplasty skin remnants.
* Healthy donors of bandages soiled with exudates from cutaneous wounds: subject consulting a plastic surgery department as part of their usual post-operative follow-up, who have given their consent for the collection of one of their dressings during their usual during their usual renewal.

For all subjects :

* Free, informed, written consent, signed by the person and the investigator no later than the day of inclusion and before any examination carried out as part of the study.
* Person affiliated or benefiting from a social security scheme

Exclusion Criteria:

EBDR patients :

* EBH with no definite diagnosis or other than EBDR intermediate, reversed or generalized
* Systemic anti-inflammatory or immunosuppressive therapy for less than one month
* Refusal of skin biopsy

Healthy controls :

* Acute or chronic systemic or cutaneous inflammatory disease at the time of sampling
* Current immunosuppressive anti-inflammatory treatment in the month prior to sampling

For all subjects:

* Persons under guardianship or curatorship, or deprived of their liberty by judicial or administrative decision
* Patients receiving State Medical Aid
* Pregnant or breast-feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with recessive dystrophic epidermolysis bullosa and healthy control patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Analysis of the cellular (PBMC) and cytokine (serum) immunological signature in the peripheral blood of EBDR subjects and healthy controls. | Up to 1 year

SECONDARY OUTCOMES:
Cellular, cytokine, and lipid immunological signatures of immune cells | Up to 1 year
  Immune cells are purified from skin biopsies and soiled dressings of EBDR patients and healthy controls. Individual data will be correlated to the severity grade of EBD.
Immunogenicity and impact of WJ-MSCs and trophoblasts | Up to 1 year
  Immunogenicity and impact of WJ-MSCs and trophoblasts on cellular, cytokine, and lipid immunological signatures, activation, and proliferation of peripheral or cutaneous immune cells from EBDR patients and healthy controls, using in-vitro models.
Immunogenicity and impact of EV/Ex | Up to 1 year
  Immunogenicity and impact of EV/Ex on cellular, cytokine, and lipid immunological signatures, activation, and proliferation of peripheral or cutaneous immune cells of EBDR patients and healthy controls, using in-vitro models.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Al-Daccak, Dr, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - Hopital Saint Louis - Service de chirurgie plastique reconstructrice et esthétique et traitement chirurgical des brûlés, Paris
  - Hopital Saint Louis - service dermatologie, Paris

IPD SHARING:
Plan to Share IPD: Undecided